CLINICAL TRIAL: NCT00651027
Title: An Open Label Study, To Evaluate The Pharmacokinetics, Safety And Toleration Of A Single Oral Dose Of Pf-00868554 In Subjects With Hepatic Impairment To Subjects With Normal Hepatic Function
Brief Title: Study To Assess The Impact Of Hepatic Impairment On The Safety, Tolerability And Pharmacokinetics Of Single-Dose 200 Mg Of PF-868554
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A8121004
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: HEPATITIS C (HCV)
MeSH Terms: conditions — Hepatitis C | interventions — filibuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: PF-868554
- B (Experimental)
  Interventions: Drug: PF-868554
- C (Experimental): 200 mg
  Interventions: Drug: PF-868554

INTERVENTIONS:
Drug: PF-868554 — 200 mg, Child-Pugh Class A
  Arms: A
Drug: PF-868554 — 200 mg, Child-Pugh Class B
  Arms: B
Drug: PF-868554 — 200 mg, healthy volunteers
  Arms: C

SUMMARY:
The metabolism of PF-00868554 is primarily mediated by CYP3A, and it is anticipated that hepatic impairment will modify PF-00868554 plasma concentrations. Hence, it is important to determine the impact of varying degrees of hepatic impairment on the pharmacokinetics, safety and toleration of 200 mg PF-00868554 administered as a single-dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or females subjects of non-childbearing potential between the ages of 18 and 62 years of age, inclusive;
* Body Mass Index (BMI) of approximately 18 to 35 kg/m2; and a total body weigh >50 kg (110 lbs);

Exclusion Criteria:

* Subjects with Class C classification (Severe - Child-Pugh Scores greater than 10);
* Severe ascites and/or pleural effusion;
* Had a transplanted kidney, heart or liver;

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
PK parameters | 8 day

SECONDARY OUTCOMES:
safety and tolerability | 8days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Miami, Florida

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8121004&StudyName=Study%20To%20Assess%20The%20Impact%20Of%20Hepatic%20Impairment%20On%20The%20Safety%2C%20Tolerability%20And%20Pharmacokinetics%20Of%20Single-Dose%20200%20Mg%20Of%20PF-868554